CLINICAL TRIAL: NCT03888729
Title: Simplifying Hepatitis C Antiviral Therapy in Rwanda for Elsewhere in the Developing World: Pangenotypic and Retreatment Study (SHARED3)
Brief Title: Simplifying HCV Treatment in Rwanda for Elsewhere in the Developing World: Pangenotypic and Retreatment Study (SHARED3)
Acronym: SHARED3
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Partners in Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PartnersIH
Record Dates: First submitted 2019-02-15; First posted 2019-03-25 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; direct-acting antiviral; Rwanda
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — velpatasvir; sofosbuvir-velpatasvir drug combination; sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of the following two groups in parallel for the duration of the study, based on treatment indication to be put on SOF/VEL or SOF/VEL/VOX:
  * sofosbubir/velpatasvir (SOF/VEL) FDC once daily for 12 weeks will be administered to HCV-infected individuals naïve to DAA therapy regimen (in this group we consider also HCV-infected individuals who have failed interferon-based therapy) who meet other eligibility criteria;
  * sofosbubir/velpatasvir /voxilaprevir (SOF/VEL/VOX) FDC once daily for 12 weeks will be administered to HCV treatment-experienced participants (i.e. HCV-infected individuals with a history of virologic failure to SOF/LDV or other DAA-containing regimen) who meet other eligibility criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HCV treatment-naïve participants (Experimental): HCV-infected individuals naïve to DAA therapy regimen; in this group we consider also HCV-infected individuals who have failed interferon-based therapy. Sofosbubir/velpatasvir (SOF/VEL) will be administered once daily for 12 weeks to eligible HCV treatment-naïve participants.
  Interventions: Drug: sofosbubir/velpatasvir
- HCV treatment-experienced participants (Experimental): HCV treatment-experienced participants, i.e.HCV-infected individuals with a history of virologic failure to SOF/LDV or other DAA-containing regimen. Sofosbubir/velpatasvir /voxilaprevir (SOF/VEL/VOX) will be administered once daily for 12 weeks to eligible HCV treatment-experienced participants
  Interventions: Drug: sofosbubir/velpatasvir/voxilaprevir

INTERVENTIONS:
Drug: sofosbubir/velpatasvir — SOF/VEL (400 mg/100 mg) FDC once daily
  Other Names: Epclusa
  Arms: HCV treatment-naïve participants
Drug: sofosbubir/velpatasvir/voxilaprevir — SOF/VEL/VOX (400 mg/100 mg/100 mg) FDC once daily
  Other Names: Vosevi
  Arms: HCV treatment-experienced participants

SUMMARY:
The main purpose of the study is to determine the antiviral efficacy and evaluate the safety and tolerability of sofosbuvir/ velpatasvir (SOF/VEL) and sofosbuvir/ velpatasvir/ voxilaprevir (SOF/VEL/VOX) used to treat individuals with chronic hepatitis C virus infection in Rwanda adults.

DETAILED DESCRIPTION:
This is an open-label single-arm study that will examine the antiviral efficacy, safety and tolerability of 12 weeks daily therapy with fixed dose combination (FDC) of SOF/VEL and SOF/VEL/VOX administered respectively in HCV-infected treatment-naïve adult participants and in HCV-infected individuals with a history of virologic failure to SOF/LDV or other DAA-containing regimen. A total of 100 participants will be enrolled in this portion of the SHARED study, labelled the "SHARED 3 study": 60 treatment-naïve participants and 40 individuals with history of virologic failure to SOF/LDV or other DAA-containing regimen

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age ≥ 18 years
* HCV RNA >1000 IU/mL at Screening
* For SOF/VEL arm, HCV treatment-naïve or interferon/ribavirin-experienced
* For SOF/VEL/VOX arm, history of virologic failure to SOF/LDV or other DAA-containing regimen as defined by a quantifiable HCV viral load any time at or after the end of HCV therapy
* Screening ultrasound excluding hepatocellular carcinoma (HCC)
* Acceptable laboratory values including:

  * Hemoglobin ≥8.0 g/dL
  * Platelet count ≥40,000/mm3
  * AST, ALT, and alkaline phosphatase ≤10 × ULN
  * Calculated creatinine clearance (CrCl) ≥30 mL/min
* General good health
* Ability to comply with the dosing instructions for study drug administration and to complete the study schedule of assessments
* If HIV-infected:

  * The participant must have completed at least 6 months of any approved HIV antiretroviral therapy (ART) before starting enrollment
  * The participant at time of screening and for at least 2 weeks prior to screening must be on ART compatible with SOF/VEL and SOF/VEL/VOX
  * Screening HIV RNA < 200 copies/mL
  * Screening CD4 T-cell count of ≥100 cells/µL
* Women of reproductive potential must have a negative urine pregnancy test at Screening and a negative urine pregnancy test at Entry prior to enrollment.

Exclusion Criteria:

* Current or history of clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage)
* Active tuberculosis
* Other clinically-significant illness (except HCV and/or HIV) or any other major medical disorder that, in the opinion of the site investigator, may interfere with participant treatment, assessment or compliance with the protocol; participants currently under evaluation for a potentially clinically-significant illness (other than HCV/HIV) are also excluded.
* Active Hepatitis B infection
* Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy
* Pregnant or nursing female
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study procedures and treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with sustained viral response 12 weeks after discontinuation of study treatment (SVR12) | After study completion (week 24)
  Antiviral efficacy of SOF/VEL FDC and SOF/VEL/VOX FDC as measured by the proportion of participants with sustained viral response 12 weeks after discontinuation of study treatment (SVR12) in Rwanda
Proportion of patients treated with SOF/VEL FDC and SOF/VEL/VOX FDC with a new grade 3 or 4 adverse event as defined by the DAIDS Scales or with premature study drug discontinuation due to an adverse event | After study completion (week 24)
  Proportion of patients treated with SOF/VEL FDC and SOF/VEL/VOX FDC with a new grade 3 or 4 adverse event as defined by the DAIDS Scales or with premature study drug discontinuation due to an adverse event

SECONDARY OUTCOMES:
Proportion of participants by HCV genotype subtypes with SVR12 after completing treatment with SOF/VEL FDC and SOF/VEL/VOX FDC | After study completion (week 24)
  Proportion of participants by HCV genotype 4 subtype with SVR12 after completing the study treatment with SOF/VEL FDC and SOF/VEL/VOX FDC
Adherence to SOF/VEL FDC and SOF/VEL/VOX FDC | After study completion (week 24)
  Proportion of participants with adequate adherence to SOF/VEL FDC and SOF/VEL/VOX FDC measured by pill count >90% of pills taken
Odds ratio for achievement of SVR12 by treatment type for the following variables: age (per 10 year increase), female sex, HIV co-infection, genotype subtype 4r, baseline HCV viral load (per 1 log increase), APRI > 1.0 | After study completion (week 24)
  Odds ratio for achievement of SVR12 by treatment type for the following variables: age (per 10 year increase), female sex, HIV co-infection, genotype subtype 4r, baseline HCV viral load (per 1 log increase), APRI > 1.0
Proportion of HIV co-infected subjects that maintain HIV-1 RNA< 200 copies/mL while on HCV treatment | After study completion (week 24)
  Proportion of HIV co-infected subjects that maintain HIV-1 RNA< 200 copies/mL while on HCV treatment, with HIV-1 RNA test performed at completion of the study treatment (week 12)
Effect of SOF/VEL FDC and SOF/VEL/VOX FDC and SVR12 on quality of life | After study completion (week 24)
  Effect of SOF/VEL FDC and SOF/VEL/VOX FDC and SVR12 on quality of life, using the MOS HIV questionnaire, with proportion of patients showing significant improvement on physical quality of life and mental quality of life from pre- to post- treatment

CONTACTS AND LOCATIONS:
Overall Officials: Neil Gupta, MD, MPH, Principal Investigator — Partners In Health; Brigham and Women's Hospital; Harvard Medical School; Fredrick Kateera, MD, PhD, Principal Investigator — Partners In Health/Inshuti Mu Buzima - Rwanda
Locations (1):
- Rwanda Military Hospital, Kigali, Rwanda

REFERENCES:
- [Result] Gupta N, Mbituyumuremyi A, Kabahizi J, Ntaganda F, Muvunyi CM, Shumbusho F, Musabeyezu E, Mukabatsinda C, Ntirenganya C, Van Nuil JI, Kateera F, Camus G, Damascene MJ, Nsanzimana S, Mukherjee J, Grant PM. Treatment of chronic hepatitis C virus infection in Rwanda with ledipasvir-sofosbuvir (SHARED): a single-arm trial. Lancet Gastroenterol Hepatol. 2019 Feb;4(2):119-126. doi: 10.1016/S2468-1253(18)30382-0. Epub 2018 Dec 11. PMID 30552056
- [Derived] Kateera F, Shumbusho F, Manirambona L, Kabihizi J, Murangwa A, Serumondo J, Makuza JD, Nsanzimana S, Muvunyi CM, Kabakambira JD, Sylvain H, Camus G, Grant PM, Gupta N. Safety and efficacy of sofosbuvir-velpatasvir to treat chronic hepatitis C virus infection in treatment-naive patients in Rwanda (SHARED-3): a single-arm trial. Lancet Gastroenterol Hepatol. 2022 Jun;7(6):533-541. doi: 10.1016/S2468-1253(21)00398-8. Epub 2022 Mar 3. PMID 35248213
- [Derived] Gupta N, Manirambona L, Shumbusho F, Kabihizi J, Murangwa A, Serumondo J, Makuza JD, Nsanzimana S, Muvunyi CM, Mukabatsinda C, Musabeyezu E, Camus G, Grant PM, Kateera F. Safety and efficacy of sofosbuvir-velpatasvir-voxilaprevir for re-treatment of chronic hepatitis C virus infection in patients with previous direct-acting antiviral treatment failure in Rwanda (SHARED-3): a single-arm trial. Lancet Gastroenterol Hepatol. 2022 Jun;7(6):542-551. doi: 10.1016/S2468-1253(21)00399-X. Epub 2022 Mar 3. PMID 35248212